CLINICAL TRIAL: NCT02773472
Title: Post-operative Electroacupuncture as Part of the Multimodal Analgesic Regimen for Laparoscopic or Robotic Colorectal Surgery
Brief Title: Electroacupuncture for Laparoscopic/ Robotic Colorectal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW15-214
Record Dates: First submitted 2015-05-27; First posted 2016-05-16 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain
Keywords: colorectal; electroacupuncture; laparoscopic surgery
MeSH Terms: conditions — Acute Pain | interventions — Electroacupuncture; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture Group (Experimental): In addition to morphine, patients will receive 4 sessions of electroacupuncture after surgery over four days, with each session lasting 30 minutes.
  Interventions: Device: electroacupuncture
- Morphine Group (Other): Neither electroacupuncture nor sham acupuncture will be given. Patient use morphine for analgesia.
  Interventions: Drug: morphine

INTERVENTIONS:
Device: electroacupuncture — The acupoints that will be stimulated are: daheng, tianshu, zhongwan, xiawan, qihai, guanuian, hegu, guchi, zusanli, sanyinjiao, gongsun. An alternating fast-slow frequency of 20Hz/6Hz will be used with an interval of 250msec. The intensity (mA) will be adjusted to a level tolerated by each individual patient.
  Arms: Electroacupuncture Group
Drug: morphine — Patient will not receive electroacupuncture. Patient will use morphine for analgesia.
  Arms: Morphine Group

SUMMARY:
A multimodal approach for management of post-operative pain is used to improve analgesia, minimize side effects, and improve recovery. Nevertheless, opioid analgesics and intravenous patient controlled analgesia remains the mainstay of postoperative analgesia after colorectal surgery. Opioids are associated with various side effects such as nausea, vomiting, sedation, dizziness, respiratory depression, urinary retention and reduced bowel movement. These side effects are unpleasant and lead to prolonged recovery.

Use of non-pharmacological analgesic techniques may improve postoperative pain control and reduce opioid consumption. Acupuncture has been used for over 3000 years in China for treatment of pain and various other conditions. Acupuncture and related techniques are simple and safe. There is evidence that acupuncture can reduce postoperative pain intensity, opioid consumption, and opioid related side effects.

DETAILED DESCRIPTION:
Procedures Patients will be approached at the pre admission clinic or in the general ward before the operation. The analgesic modalities will be explained and the patient will be recruited into the study if s/he agrees. The patient will subsequently be randomized into one of two groups. Patients in the first group (M) will receive intraoperative morphine, local wound infiltration with local anaesthetic, paracetamol, cyclooxygenase-2 (COX-2) inhibitor and postoperative patient controlled analgesic (PCA) morphine. Patients in the second group (E) will receive postoperative electroacupuncture in addition to intraoperative morphine, local wound infiltration with local anaesthetic, COX-2 inhibitor, paracetamol and postoperative PCA morphine.

Randomization and blinding Patients recruited for laparoscopic colonic and rectal surgery will be stratified in randomization. To ensure all groups have equal sample size, each randomization will be based on using 10 blocks of 10 patients for each type of operation (colonic and rectal). A computer generated random sequence will be used to select the allocation order.

This is a single blinded randomized control trial. Blinding will not be done for the patients. The investigator assessing the patients for data collection after the operation will be blinded.

Analgesic modalities and pain assessment Group E In addition to the standard protocol applied to patients in group M, patients in the electroacupuncture group (E) will receive 4 sessions of electroacupuncture after surgery over four days, with each session lasting 30 minutes. The first session will start 3 hours after surgery on post op day 0. Subsequently, patients will receive 1 sessions each morning on post op days 1, 2, and 3. The acupoints that will be stimulated are: daheng, tianshu, zhongwan, xiawan, qihai, guanyuan, hegu, quchi, zusanli, sanyinjiao, gongsun. An alternating fast-slow frequency of 20Hz/6Hz will be used with an interval of 250msec. The intensity (mA) will be adjusted to a level tolerated by each individual patient. Electroacupuncture will be performed by qualified acupuncturists from the School of Chinese Medicine, The University of Hong Kong.

Group M Patients in group M will receive intravenous morphine, paracetamol, COX-2 inhibitor, local wound infiltration with local anaesthetic and post operative PCA morphine only as mentioned above. Neither electroacupuncture nor sham acupuncture will be given.

Postoperative care and assessment Early mobilization is encouraged after operation. Patients will be put on fluid diet on postoperative day 0.

Postoperative assessments such as gastrointestinal function (bowel sound, flatus, bowel opening), occurrences of postoperative complications, and suitability for discharge (good pain control, ambulation, normal bowel function, ability to eat properly without vomiting or abdominal distention) would be performed by the surgical team.

Pain control using the numerical rating scale (NRS) scale from 0-10 and patient satisfaction with analgesia will be assessed upon discharge.

Blood sampling In order to determine the plasma concentrations of adenosine, encephalin, beta-endorphin, dynorphin and alpha-endomorphin, and methylation status and gene expression of mu-, delta- and kappa-opioid receptors, 10 mls of blood will be drawn (4 mls into Ethylenediaminetetraacetic acid (EDTA) and 6 mls into heparinised blood collection tubes) at the following time-points in all subjects: Prior to first acupuncture session, prior to second acupuncture session, prior to 4th acupuncture session and prior to 6th acupuncture session.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists adopted physical status classification system (ASA) I to III
* Age 18 to 80 years old
* Scheduled for elective laparoscopic/ robotic colonic or upper rectal resection in Queen Mary hospital.

Exclusion Criteria:

* Open colorectal surgery
* Extended resection involving other organs such as liver and urinary bladder
* Known drug allergy to alpha-2 agonists, opioids, non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2 inhibitors, paracetamol, or sulphonamides
* Alcohol or drug abuse
* Known history of pulmonary embolism or deep vein thrombosis
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Impaired hepatic function, defined as preoperative serum albumin level less than 30g/L
* Impaired or retarded mental state
* Not self-ambulatory before operation
* Difficulties in using patient-controlled analgesia
* Body Mass Index > 35kg/m2
* Pregnancy
* Local infection
* Abdominal wound
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Acute pain | at postoperative day 3
  Severity of postoperative pain will be assessed using numerical rating scale

SECONDARY OUTCOMES:
Chronic pain | at postoperative 3 months
  Presence of persistent pain will be assessed using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No